CLINICAL TRIAL: NCT00641186
Title: A Phase II, Eight Week, Multi-Center, Open Label Trial of Xyrem(R) (Sodium Oxybate) for Excessive Daytime Sleepiness and Nocturnal Sleep Disturbance in Patients With Mild to Moderate Parkinson's Disease
Brief Title: Trial of Xyrem for Excessive Daytime Sleepiness and Sleep Disturbance in Parkinson's Disease (PD)
Acronym: Xyrem
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Joseph Jankovic, Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-16378
Record Dates: First submitted 2008-03-18; First posted 2008-03-24 (Estimated); Results first posted 2022-09-28 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-09

CONDITIONS: Parkinson Disease
Keywords: excessive daytime somnolence; Parkinson disease; sleep disturbance
MeSH Terms: conditions — Parkinson Disease; Disorders of Excessive Somnolence; Parasomnias | interventions — Sodium Oxybate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Xyrem in Parkinson disease (Experimental): sodium oxybate 4.5 to 9.0 gms per night
  Interventions: Drug: sodium oxybate

INTERVENTIONS:
Drug: sodium oxybate — 4.5 to 9.0 grams per night
  Other Names: Xyrem

SUMMARY:
This clinical trial is designed to evaluate the safety and potential efficacy of Xyrem for the treatment of excessive daytime sleepiness (EDS) and nocturnal sleep disturbance in patients with mild to moderate Parkinson's Disease (PD).

DETAILED DESCRIPTION:
Inclusion required an Epworth Sleepiness Scale (ESS) score greater than 10 and any subjective nocturnal sleep concern, usually insomnia. An acclimation and screening polysomnogram was performed to exclude subjects with sleepdisordered breathing. The following evening, subjects underwent another polysomnogram, followed by an evaluation with the Unified Parkinson Disease Rating Scale (UPDRS) while practically defined off ("off") PD medications, ESS (primary efficacy point), Pittsburgh Sleep Quality Inventory, and Fatigue Severity Scale. Subjects then started sodium oxybate therapy, which was titrated from 3 to 9 g per night in split doses (at bedtime and 4 hours later) across 6 weeks, and returned for subjective sleep assessments. They then returned at 12 weeks after initiating therapy for a third polysomnogram, an offmedication UPDRS evaluation, and subjective sleep assessments. Data are expressed as mean (SD).

ELIGIBILITY:
Inclusion Criteria:

* Male or female with a diagnosis of idiopathic PD.
* Age between 30 and 75, inclusive. -Hoehn & Yahr Stage 1.5 - 4.0 in the practically defined medication "OFF". -
* History > 2 months of excessive daytime sleepiness confirmed at baseline/screening by an Epworth Sleepiness Scale score of > 10.
* History > 2 months of nocturnal sleep disturbances consisting of insomnia, fragmented sleep and/or non-restorative sleep.
* Folstein Mini-Mental State Exam score of > 24.
* Birth control for sexually active women of childbearing potential (e.g. abstinence, hormonal contraception, barrier method, intrauterine device).
* Evidence of a personally signed and dated informed consent form document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the trial.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, and other study procedures.
* Stable dose of medications, defined as no change in dose or regimen of medications for at least 3 months prior to Screen Visit.

Exclusion Criteria:

* Known idiopathic sleep pathology: sleep apnea and narcolepsy.
* Serious co-morbid disease --Atypical parkinsonism (e.g., Parkinson "plus" syndrome, secondary Parkinson's syndrome). --Significant neurological symptoms not accounted for by PD. --Significant psychiatric symptoms or dementia.
* Sexually active women of childbearing potential without adequate form of birth control.
* Pregnancy or lactation.
* Mini-mental status examination of < 25.
* Participation in another clinical trial of another investigational agent or device within the previous 60 days.
* Current abuse of alcohol or drugs.
* Active or prior malignancy other than cutaneous basal cell carcinoma or in situ carcinoma of the uterine cervix.
* Known hypersensitivity to sodium oxybate or other constituents of the product.
* Any medical conditions that are contraindications to the use of sodium oxybate or significant hepatic impairment.
* Patients being treated with sedative hypnotic agents or other central nervous system (CNS) depressants.
* Subjects taking warfarin.
* Patients with succinic semialdehyde dehydrogenase deficiency.
* Subjects who, in the opinion of the investigator, are not able to comply with the requirements of the study.
* Any other condition that, in the investigator's opinion, would cause a significant hazard to the subject.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-09; Primary Completion 2008-07 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William G Ondo, MD, Principal Investigator — Baylor College of Medicine

REFERENCES:
- [Background] Ondo WG, Perkins T, Swick T, Hull KL Jr, Jimenez JE, Garris TS, Pardi D. Sodium oxybate for excessive daytime sleepiness in Parkinson disease: an open-label polysomnographic study. Arch Neurol. 2008 Oct;65(10):1337-40. doi: 10.1001/archneur.65.10.1337. PMID 18852348

RESULTS

PARTICIPANT FLOW:
Groups:
- Trial of Xyrem for Excessive Daytime Sleepiness and Sleep Dist: Xyrem arm, single arm study for excessive daytime sleepiness and sleep disturbance in PD
Period: Overall Study
Arm/Group | Trial of Xyrem for Excessive Daytime Sleepiness and Sleep Dist
Started | 30
Completed | 27
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Population: These participants were in the Xyrem arm, single arm study for excessive daytime sleepiness and sleep disturbance in PD
Groups:
- Treatment Group: Active treatment group with Xyrem in PD
Arm/Group | Treatment Group
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Sleep and Fatigue
Description: Sleep and Fatigue was measured using the following scales before and after sodium oxybate therapy Scales used to measure sleep and fatigue: Epworth Sleepiness Scale (ESS) where score ranges from 0-24 where 0 = no sleep problems and 24 = excessive sleep problems that should seek medical attention; Fatigue Severity Scale (FSS) where the score ranges from 9-36 where 9 = no fatigue and 36 = severe fatigue; Pittsburgh Sleep Quality Inventory (PSQI) where the score ranges from 0-21 where any score greater than 5 indicates a great sleep disturbance; 36-Item Short Form Health Survey (SF-36) where the score ranges 0-100 where 0 = the worst health status and 100 = the best health status. * Findings are reported for 28 subjects. The Full Range values reported reflect the measured minimum and maximum values.
Time Frame: 8 weeks
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Trial of Xyrem for Excessive Daytime Sleepiness and Sleep Disturbance: Xyrem arm, single arm study for excessive sleep disturbance in PD
Arm/Group | Trial of Xyrem for Excessive Daytime Sleepiness and Sleep Disturbance
Number analyzed (Participants) | 28
units on a scale
  Before Sodium Oxybate Therapy (baseline) ESS | 15.6 [0 to 24]
  After Sodium Oxybate Therapy (8 weeks) ESS | 9.0 [0 to 24]
  Before Sodium Oxybate Therapy (baseline) PSQI | 10.9 [0 to 21]
  After Sodium Oxybate Therapy (8 weeks) PSQI | 6.6 [0 to 21]
  Before Sodium Oxybate Therapy (baseline) FSS | 32.9 [9 to 36]
  After Sodium Oxybate Therapy (8 weeks) FSS | 26.3 [9 to 36]
  Before Sodium Oxybate Therapy (baseline) SF-36 | 95.7 [0 to 100]
  After Sodium Oxybate Therapy (8 weeks) SF-36 | 92.3 [0 to 100]

2. Secondary Outcome: Polysomnography (PSG)
Description: Polysomnography, also called a sleep study, is a comprehensive test used to diagnose sleep disorders. The minimum score would be 0, the maximum score would be 30. A score of 0 - 4 = normal sleep, a score of 5 - 14 = a mild level of sleep disturbance, a score of 15 - 30 is moderate level of sleep disturbance and a score of 30 is severe sleep disturbance.
Time Frame: 8 weeks
Population: A polysomnography was done before and after therapy as a secondary measure. The results are below.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Trial of Xyrem for Excessive Daytime Sleepiness and Sleep Disturbance
Number analyzed (Participants) | 27
units on a scale
  Mean Polysomnography Before Therapy | 7 [0 to 14]
  Mean Polysomnography After Therapy | 13 [0 to 30]

ADVERSE EVENTS:
Time Frame: Screening through follow-up for a total duration 56 days.
Description: Any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, and which does not necessarily have a causal relationship with that treatment.
Groups:
- All Subjects: Adverse events probably or definitely related to the drug included:
  nocturia/enuresis (n=3), dizziness and nausea (n=1), dizziness with daytime sleepiness reduced alertness (n = 1), dizziness with rebound morning tremor (n=1).
  Additional adverse events that were considered not related to the study drug included: constipation (n=1),1 delusions (n=1), and, in a single subject, bradycardia, anxiety, depression, and edema.
  Twenty-one of 30 subjects (70%) reported no adverse events.
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 9/30
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=30)
enuresis (Renal and urinary disorders) | 3 (3)
rebounding morning tremor (Nervous system disorders) | 1 (1)
dizziness (General disorders) | 3 (3)
daytime sleepiness (General disorders) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1)
delusions (Psychiatric disorders) | 1 (1)
bradycardia (General disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
depression (Psychiatric disorders) | 1 (1)
edema (Blood and lymphatic system disorders) | 1 (1)
nausea (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No